CLINICAL TRIAL: NCT00893620
Title: Zenith(R) Connection Endovascular Covered Stent Clinical Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to less than expected enrollment rates, Cook has reevaluated the need for this clinical study.
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-007; 370020, BVCT
Record Dates: First submitted 2009-04-27; First posted 2009-05-06 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2012-01

CONDITIONS: Aorto-iliac Aneurysms; Iliac Aneurysms
Keywords: iliac aneurysm; endovascular repair
MeSH Terms: conditions — Iliac Aneurysm

ARMS (1):
- 1 (Other): Treatment
  Interventions: Device: Zenith(R) Connection Endovascular Covered Stent with the Zenith® Branch Endovascular Graft-Iliac Bifurcation and Zenith Flex(R) AAA Endovascular Graft

INTERVENTIONS:
Device: Zenith(R) Connection Endovascular Covered Stent with the Zenith® Branch Endovascular Graft-Iliac Bifurcation and Zenith Flex(R) AAA Endovascular Graft — These devices will be used in patients with an unsuitable distal sealing site for the standard Zenith(R) iliac leg component proximal to the common iliac bifurcation to maintain internal iliac artery patency with endovascular aneurysm repair.
  Other Names: Zenith(R) Connection Endovascular Covered Stent

SUMMARY:
The Zenith(R) Connection Endovascular Covered Stent Clinical Study is a clinical investigation to study the safety and performance of the Zenith(R) Connection Endovascular Covered Stent in conjunction with the Zenith(R) Branch Endovascular Graft-Iliac Bifurcation in the treatment of aorto-iliac and iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* An aortoiliac or iliac aneurysm of appropriate size
* Unsuitable distal sealing site for a traditional Zenith® iliac leg graft within the common iliac artery

Exclusion Criteria:

* Less than 18 years of age
* Inability or refusal to give informed consent
* Disease considerations that would compromise patient safety or study outcomes
* Unsuitable arterial anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Deployment and procedural outcome | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lee, MD, Principal Investigator — Christine E. Lynn Heart and Vascular Institute
Locations (4):
- Germany (2):
  - St. Bonifatius Hospital GmbH, Lingen
  - St. Franziskus Hospital, Münster
- Queen Mary Hospital, Hong Kong, Hong Kong
- Manchester Royal Infirmary, Manchester, United Kingdom